CLINICAL TRIAL: NCT04043936
Title: Increasing Connection to Care Among Military Service Members at Elevated Suicide Risk: A Randomized Controlled Trial of a Web-Based Intervention
Brief Title: Increasing Help-Seeking in Military Service Members
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida State University (Other)
Collaborators: Military Suicide Research Consortium (Other)
Responsible Party: Principal Investigator, Thomas Joiner, The Robert O. Lawton Professor in the Department of Psychology, Florida State University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Health Services Research
Other Study IDs: 043716
Record Dates: First submitted 2019-08-01; First posted 2019-08-02 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2023-04

CONDITIONS: Military Service Members at Elevated Suicide Risk
Keywords: suicide prevention; reducing stigma
MeSH Terms: conditions — Suicide Prevention

STUDY DESIGN:
Intervention Model Description: Participants will be placed in one of three groups (Cognitive Bias Modification Intervention for Help-Seeking Stigma (CBM-HS) condition, the Cognitive Bias Modification (CBM-Placebo) condition, or the Self-Directed Psychoeducation condition [comparison condition]). Participants will then complete 5 additional virtual study visits (3 intervention weeks, 1 post-treatment, 1 two-month follow-up); these study visits will occur through a web-based platform. Self-report measures will be administered at enrollment/baseline, mid-intervention, post-intervention, and two-month follow-up.
Who Masked: Participant
Masking Description: Participant will be in the Cognitive Bias Modification Intervention for Help-Seeking Stigma (CBM-HS) condition (intervention condition), the Cognitive Bias Modification (CBM-Placebo) condition (placebo condition), or the Self-Directed Psychoeducation condition (comparison condition).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cognitive Bias Modification for Help-Seeking Stigma (CBM-HS) (Experimental): CBM-HS is a 15-minute web-based intervention designed to alter maladaptive cognitions related to mental health help-seeking. In this task, individuals are presented with a series of statements regarding beliefs about using behavioral health services. Individuals then select "True" or "False" in response to each statement. Incorrect responses (i.e., demonstrating help-seeking stigma) are followed by corrective feedback. Conversely, correct responses (i.e., promoting help-seeking) are positively reinforced. Participants in this condition will complete three separate 15-minute CBM-HS sessions.
  Interventions: Behavioral: Cognitive Bias Modification Intervention for Help-Seeking Stigma
- Placebo Cognitive Bias Modification (Sham Comparator): Participants randomized to this condition will complete a CBM task with a neutral stimuli. The duration of the CBM-Placebo task will be comparable to the duration of the CBM-HS task (i.e., three 15-minute sessions).
  Interventions: Behavioral: Placebo Cognitive Bias Modification (CBM-Placebo)
- Self-Directed Psychoeducation (Active Comparator): Participants randomized to this condition will review psychoeducation on mental health literacy, mental illness stigma, and treatment options. Readings will be compiled from resources available in the public domain. The duration will be comparable to the duration of study tasks for individuals in the CBM-HS study condition (i.e., three 15-minute sessions).
  Interventions: Behavioral: Self-Directed Psychoeducation

INTERVENTIONS:
Behavioral: Cognitive Bias Modification Intervention for Help-Seeking Stigma — Cognitive bias modification (CBM) is an intervention designed to target stigma-related cognitions among individuals at elevated suicide risk not currently engaged in behavioral health treatment. It involves the completion of brief, web-based tasks in which participants are presented with a series of stimuli (e.g., words, sentences) and trained to respond to those stimuli in a manner that is positive or neutral, rather than negative and unhelpful. Consistent with the theoretical rationale for Cognitive Behavioral Therapy, CBM interventions function by reshaping negative cognitions. Repeated reinforcement of adaptive cognitions enhances functioning and reduces distress.
  Other Names: CBM-HS
  Arms: Cognitive Bias Modification for Help-Seeking Stigma (CBM-HS)
Behavioral: Placebo Cognitive Bias Modification (CBM-Placebo) — Cognitive bias modification (CBM) is an intervention designed to target stigma-related cognitions among individuals at elevated suicide risk not currently engaged in behavioral health treatment. It involves the completion of brief, web-based tasks in which participants are presented with a series of stimuli (e.g., words, sentences) and trained to respond to those stimuli in a manner that is positive or neutral, rather than negative and unhelpful. Consistent with the theoretical rationale for Cognitive Behavioral Therapy, CBM interventions function by reshaping negative cognitions. Repeated reinforcement of adaptive cognitions enhances functioning and reduces distress.
  Arms: Placebo Cognitive Bias Modification
Behavioral: Self-Directed Psychoeducation — Material presented with information on mental health literacy, mental health stigma, & treatment options. This is based on the idea that increasing knowledge about psychiatric symptoms and treatment options encourages help-seeking behavior and engagement.
  Arms: Self-Directed Psychoeducation

SUMMARY:
There is sufficient evidence that military service members markedly underutilize behavioral health care services, in part, due to stigma. This study proposes to examine a novel application of a cognitive bias modification (CBM) intervention designed to target stigma-related cognitions among service members at elevated suicide risk not currently engaged in behavioral health treatment.

DETAILED DESCRIPTION:
This study proposes to examine a novel application of a cognitive bias modification (CBM) intervention designed to target stigma-related cognitions among service members at elevated suicide risk not currently engaged in behavioral health treatment. Interventions that leverage CBM principles involve the completion of brief, web-based tasks in which participants are presented with a series of stimuli (e.g., words, sentences) and trained to respond to those stimuli in a manner that is positive or neutral, rather than negative and unhelpful. Consistent with the theoretical rationale for Cognitive Behavioral Therapy, CBM interventions function by reshaping negative cognitions. Repeated reinforcement of adaptive cognitions enhances functioning and reduces distress. CBM interventions have efficacy in reducing maladaptive cognitions across a range of psychiatric symptoms. However, limited data exist regarding the use of CBM to target help-seeking stigma cognitions.

ELIGIBILITY:
Inclusion Criteria:

* current active duty U.S. military service member
* lifetime history of suicidal ideation per a self-report version of the SITBI-SF and/or
* current elevated suicide risk factors (i.e., screening positive for clinically significant suicidal ideation [DSI-SS Total Score > 2], depression [PHQ-9 Total Score > 14], anxiety [GAD-7 Total Score > 9], PTSD [PCL-5 Total Score > 32], alcohol use [AUDIT-C Total Score > 3 for men and > 2 for women], and/or anger [DARS Total Score > 22])
* no current behavioral health service use (i.e., ongoing care with a provider to receive psychiatric medications, therapy, and/or counseling)

Exclusion Criteria:

* unable to provide informed consent
* lack of Internet access via a computer, tablet, and/or mobile phone
* scheduled to be stationed outside the continental U.S. any time during the 11 weeks following study enrollment (i.e., during the study period)
* imminent suicide risk (i.e., suicide risk warranting hospitalization) based on the Joiner et al. and Chu et al. Decision Tree Framework.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2020-04-19 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Perceived Stigma and Barriers to Care for Psychological Problems Scale (PS) | 2-Month Follow-up
  The 11-item PS measures the extent to which various concerns might affect an individual's decision to seek psychiatric treatment. Items are rated on a 5-point scale; higher scores (range: 11-55) indicate greater perceived barriers to care. The PS has been used extensively in military populations and has exhibited acceptable to good internal consistency.
Readiness to Change | 2-Month Follow-up
  Consistent with past research, we will use an adaptation of the Readiness to Change Scale to assess readiness to engage in help-seeking behaviors. Responses to each of the 6 items are anchored on an 11-point scale, with higher scores (range: 0-60) indicating greater readiness to engage in behavioral health care. Past research using this approach has yielded good internal consistency.
Self-Stigma of Seeking Help (SSOSH) | 2-Month Follow-up
  The SSOSH is a 10-item measure of help-seeking stigma. Responses are rated on a 5-point scale; higher scores (range: 0-50) reflect greater self-stigma associated with seeking help. The scale has demonstrated strong reliability and validity, and it differentiates between young adults who do and do not seek help for mental health problems.
World Mental Health Composite International Diagnostic Interview (WMH-CIDI) | 2-Month Follow-up
  A self-report version of the WMH-CIDI Services subscale will be utilized to assess the presence/absence of specific structural and attitudinal barriers to care. This WMH-CIDI has been used extensively among adult community samples, including among individuals at elevated suicide risk.
Client Satisfaction Questionnaire-8 (CSQ-8) | 2-Month Follow-up
  The CSQ-8 is an 8-item self-report measure that assesses client satisfaction with services, including mental health care services (range: 8-32). The CSQ-8 has demonstrated strong psychometric properties, including among psychotherapy patients.
Intervention Acceptability and Feasibility Questionnaire | 2-Month Follow-up
  Acceptability and feasibility will be measured using recruitment and retention rates and open-ended treatment satisfaction questions administered to participants at post-treatment (e.g., "What aspects of the intervention could be improved?").

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Florida State University, Tallahassee, Florida
  - Naval Medical Center Portsmouth, Portsmouth, Virginia

IPD SHARING:
Plan to Share IPD: No